CLINICAL TRIAL: NCT00914706
Title: Challenging the Ontario Diabetes Care Quality Gap: Evaluation and Long-Term Cost-Utility Analysis of Using a Chronic Disease Management System (CDMS) in Primary Health Care Practices in Ontario (ODIAC-CDMS): A Prospective, Observational, Comparative Study of the Effect of a CDMS on Diabetes Care Within Multidisciplinary Primary Care Practices in Ontario.
Brief Title: A Study of the Effect of a Chronic Disease Management System on Diabetes Care Within Multidisciplinary Primary Care Practices in Ontario
Status: Completed | Type: Observational
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Ron Goeree, Director, PATH Research Institute, St. Joseph's Healthcare Hamilton
Other Study IDs: FEEAP-D0014a-2009-PTL
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: P-PROMPT — P-PROMPT is a web-based chronic disease management system. The system will help to ensure that all patients have up-to-date laboratory monitoring and visits as recommended by the Canadian Diabetes Association Guidelines.

SUMMARY:
The purpose of this study is to evaluate the impact of using a web-based (P-PROMPT) chronic disease management system (CDMS) by primary care practitioners and their team members and on their care for patients with diabetes. The system will help to ensure that all patients have up-to-date laboratory monitoring and visits as recommended by the Canadian Diabetes Association Guidelines. The hypothesis is that the use of a CDMS in Ontario primary care practices, as a part of the routine clinical management of diabetes patients, can improve monitoring frequency of A1C, blood pressure (BP) and cholesterol levels. The results of this study will serve as a benchmark for the utilization of chronic disease management software tools in primary care diabetes management for patients in Ontario, establishing and providing evidence to inform decision-makers. If the results are favorable towards CDMS interventions for the management of diabetes, potential expansion and availability of these types of programs may be possible for other chronic diseases.

DETAILED DESCRIPTION:
Practice Guidelines recommend that patients with chronic diseases should be monitored with specified clinical measurements each with regular repeats at different specified time intervals or on specified conditions. It is virtually impossible for health care providers to adhere consistently to guidelines and to do so sustainability as well as equitably for "most if not all" of their patients with diabetes. Ontario Health Technology Advisory Committee (OHTAC) has requested the following study. Aggregate monthly primary care practice level data will form the basis of the analysis. Primary care practitioners in Ontario will be enrolled. Differences in 1-year outcome measures within will be performed. Baseline, 2 month, 6 month and 12 month site team member surveys will be completed. Using patient level data from each site, a cost-utility analysis will be conducted. Six aspects related to the use of the CDMS will be examined.

1. Change in proportion of the patients in whom monitoring frequency is up to date for A1C, blood pressure and cholesterol.
2. Change in proportion of patients who are well controlled with A1C < 0.07, blood pressure < 130/80 and LDL-cholesterol < 2.0.
3. Change from baseline across sites in the percentage of patients with an up-to-date foot exam, retinopathy screening, use of angiotensin converting enzyme inhibitors (ACEi) or angiotensin II receptor blockers (ARB) and documentation of self-management goals.
4. Site questionnaires.
5. Changes in physician MOHLTC diabetes incentive billings.
6. Long-term cost-utility of the use of the CDMS.

ELIGIBILITY:
Inclusion Criteria:

* Ontario primary care practitioners able to provide a list of patients within their practice.
* High-speed internet access in the practice environment or willingness to obtain high-speed internet access.
* Physicians willing to use the CDMS or already using it currently.

Exclusion Criteria:

* Ontario primary care practitioners involved in the QIIP Learning Collaboratives who are practicing in one of the following local health integration networks:

  * LHIN 2 South West
  * LHIN 7 Toronto Central
  * LHIN 11 Champlain AND
  * LHIN 14 North West so as to not interfere with other Provincial diabetes initiatives.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The unit of evaluation or cluster for this study will be individual primary care practitioners. The study will analyze aggregate practice level data from all rostered diabetes patients within each practice. Between 33 and 61 primary care practitioners with a total number of patients with diabetes across all practices of 2,376 from across Ontario will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in monitoring frequency | 1 year
  Change in proportion of patients, with up-to-date monitoring of A1C (6 months), blood pressure (annually) and cholesterol (6 months) in practices using a CDMS for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ron Goeree, Principal Investigator — St. Joseph's Healthcare Hamilton/McMaster University
Locations (6):
- Canada (6):
  - Brockville Family Health Team, Brockcillw, Ontario
  - Delhi Family Health Team, Delhi, Ontario
  - Summerville Family Health Team, Etobicoke, Ontario
  - Harrow Health Centre, Harrow, Ontario
  - Leamington and Area Family Health Team, Lemington, Ontario
  - Sherbourne Family Health Team, Toronto, Ontario